CLINICAL TRIAL: NCT06267118
Title: A Randomized Controlled Trial on the Comparative Efficacy of Hypertonic Saline vs Adrenaline Nebulization in Acute Bronchiolitis in Children
Brief Title: Comparative Efficacy of Hypertonic Saline vs Adrenaline Nebulization in Acute Bronchiolitis
Acronym: children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Syed Qamar Zaman, Assistant Professor & Head of Pediatrics Department, Combined Military Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Treatment of Bronchiolitis
Record Dates: First submitted 2024-01-07; First posted 2024-02-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Acute Bronchiolitis Due to Respiratory Syncytial Virus
Keywords: Wood-Downes Clinical scoring System
MeSH Terms: interventions — Saline Solution, Hypertonic; Epinephrine

STUDY DESIGN:
Intervention Model Description: Patients with acute bronchiolitis after informed written consent will be divided into two groups randomly. Group I will be nebulized with adrenaline every 6 hours and group II will nebulized with hypertonic saline every 6 hours. After 24 hours and 48 hours of nebulization, WDF score will be recorded by measuring respiratory rate, heart rate, chest retractions, chest auscultation findings and SPO₂ levels. Researcher will record all data on a specified Performa.
Who Masked: Participant, Care Provider
Masking Description: Investigator will make all the protocol and research Performa. Drugs will already be prepared for nebulization and labelled by investigator. Researcher /care provider will nebulize the patients of both groups randomly and record the results accordingly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypertonic saline nebulization group (Active Comparator): First group of patients diagnosed as acute bronchiolitis will be nebulized with hypertonic saline every 6 hours and data will be recorded on a Performa
  Interventions: Drug: Hypertonic Saline Solution, 1 Ml
- Adrenaline nebulization group (Active Comparator): Second group of patients will be nebulized with adrenaline every 6 hours and data will be recorded on a Performa
  Interventions: Drug: Adrenaline

INTERVENTIONS:
Drug: Hypertonic Saline Solution, 1 Ml — Dilute 0.3 ml hypertonic saline with 3 ml normal saline for nebulization
  Other Names: Drug A
  Arms: Hypertonic saline nebulization group
Drug: Adrenaline — dilute 0.3 ml adrenaline with 3 ml normal saline for nebulization
  Other Names: Drug B
  Arms: Adrenaline nebulization group

SUMMARY:
The goal of this clinical trial is to compare the efficacy of hypertonic saline nebulization with adrenaline nebulization in the treatment of acute bronchiolitis in children. Main aim is to evaluate the following in both group of patients

1. Improvement in Wood-Downes clinical score (WDF score) in bronchiolitis
2. Length of Hospitalization

DETAILED DESCRIPTION:
This is a double-blind clinical trial that will include all admitted patients with acute bronchiolitis, meeting inclusion criteria, admitted in Pediatrics department Combined Military Hospital Nowshera. Patients will be divided into two groups randomly. Group I patients will be nebulized with drug adrenaline every 6 hours and group II patients will be nebulized with hypertonic saline every 6 hours. After 24 hours and 48 hours of nebulization, researchers will record WDF score by measuring respiratory rate, heart rate, chest retractions, chest auscultation findings and SPO₂ levels. All data will be recorded on a research Performa including length of hospital stay. Data will be entered on SPSS to calculate results. Independent sample t-test was used to measure the effect of two drugs on the length of hospital stay and improvement of respiratory score with a 95% confidence interval. P value less than 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted in PICU with acute bronchiolitis

Exclusion Criteria:

* children with co-exiting illnesses like

  1. Congenital Heart Disease
  2. Immunodeficiency
  3. other Infectious disease like Meningitis, encephalitis, Pneumonia, TORCH
  4. Kidneys or liver problem
  5. Seizures

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Wood-Downes-Ferres clinical score calculation | at 24 and 48 hours of treatment
  A score of 0-3 mild, 4-6 moderately ill, >6 severely ill

SECONDARY OUTCOMES:
total length of hospitalization | less than 7 days, 7-10 days, 10-14 days
  less than 1 week, more than 1 week,

CONTACTS AND LOCATIONS:
Overall Officials: Prof Shahid Mahmud, Study Director — Military Hospital Rawalpindi
Locations (1):
- Combined Military Hospital, Nowshera, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
After informed consent of participants and ethical committee approval, it will be shared.

REFERENCES:
- [Result] Piedimonte G, Perez MK. Respiratory syncytial virus infection and bronchiolitis. Pediatr Rev. 2014 Dec;35(12):519-30. doi: 10.1542/pir.35-12-519. No abstract available. PMID 25452661
- [Result] Anil AB, Anil M, Saglam AB, Cetin N, Bal A, Aksu N. High volume normal saline alone is as effective as nebulized salbutamol-normal saline, epinephrine-normal saline, and 3% saline in mild bronchiolitis. Pediatr Pulmonol. 2010 Jan;45(1):41-7. doi: 10.1002/ppul.21108. PMID 19953579
- [Result] Florin TA, Plint AC, Zorc JJ. Viral bronchiolitis. Lancet. 2017 Jan 14;389(10065):211-224. doi: 10.1016/S0140-6736(16)30951-5. Epub 2016 Aug 20. PMID 27549684
- [Result] Grewal S, Ali S, McConnell DW, Vandermeer B, Klassen TP. A randomized trial of nebulized 3% hypertonic saline with epinephrine in the treatment of acute bronchiolitis in the emergency department. Arch Pediatr Adolesc Med. 2009 Nov;163(11):1007-12. doi: 10.1001/archpediatrics.2009.196. PMID 19884591
- [Result] Zhang L, Mendoza-Sassi RA, Wainwright C, Klassen TP. Nebulised hypertonic saline solution for acute bronchiolitis in infants. Cochrane Database Syst Rev. 2017 Dec 21;12(12):CD006458. doi: 10.1002/14651858.CD006458.pub4. PMID 29265171
- [Result] Hariprakash S, Alexander J, Carroll W, Ramesh P, Randell T, Turnbull F, Lenney W. Randomized controlled trial of nebulized adrenaline in acute bronchiolitis. Pediatr Allergy Immunol. 2003 Apr;14(2):134-9. doi: 10.1034/j.1399-3038.2003.00014.x. PMID 12675760
- [Result] Fretzayas A, Moustaki M. Etiology and clinical features of viral bronchiolitis in infancy. World J Pediatr. 2017 Aug;13(4):293-299. doi: 10.1007/s12519-017-0031-8. Epub 2017 May 4. PMID 28470580
- See also: RCTnebulized epinephrine versus nebulized hypertonic saline in infants with acute bronchiolitis — https://www.ijpediatrics.com/index.php/ijcp/article/view/4218
- See also: Viral bronchiolitis in children: A common condition with few therapeutic options — http://doi.org/10.1016/j.earlhumdev.2013.07.016